CLINICAL TRIAL: NCT07390448
Title: A Comparative Study Between Ultrasound Guided Combined Rhomboid Intercostal and Sub- Serratus Plane Blocks and Erector Spinae Plane Block as Perioperative Analgesia in Mastectomy Surgeries in Cancer Breast Patients
Brief Title: Rhomboid Intercostal Sub-serratus Plane Blocks and Erector Spinae Plane Block in Mastectomy Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ayman Sharawy Abdel Rahman Aboul Nasr, Principal investigator, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AP2512-501-144-205
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: erector spinae plane block; Rhomboid Intercostal and Sub-serratus Plane Blocks; ultra sound
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided Rhomboid intercostal block sub-serratus plane block (RISS). (Active Comparator): With the patient in the lateral decubitus position, a rhomboid intercostal block will be performed under ultrasound guidance using a linear probe (6-12 MHz). The transducer will be positioned medial to the scapular border to obtain an oblique sagittal view. A 17G Tuohy needle will be advanced in-plane from a superomedial to an inferolateral direction through the trapezius and rhomboid major muscles, and 10 mL of 0.25% bupivacaine will be injected at the T5-T6 level. The probe will then be moved caudally and laterally to identify the plane between the serratus anterior and external intercostal muscles for a sub-serratus block at T6-T9. Using the same skin entry point, the needle will be redirected caudolaterally, and 15 mL of 0.25% bupivacaine will be administered superficial to the intercostal muscles.
  Interventions: Procedure: Ultrasound Guided Combined Rhomboid Intercostal Sub-serratus Plane Blocks
- Ultrasound guided Erector spinae plane block (ESPB) (Active Comparator): The patient will be placed in sitting position. The spine will be palpated from C7 downward to T5 and point will be marked to identify the spinous process. After ensuring skin asepsis, the high frequency (5-13 MHz) linear probe of ultrasound machine (Sonosite, Bothwell, USA) will be placed in a sterile sheath 3 cm lateral to the T5 spinous process. The three muscles from outward will be recognized: trapezius, rhomboidus major, and erector spinae muscle. An 18-gauge Tuohy needle will be inserted using an in-plane superior to inferior approach to place the tip into fascial plane on the deep (anterior) aspect of erector spinae muscle. The location of the needle tip was confirmed by visible fluid spread below erector spinae muscle off the bony shadow of the transverse process. A total of 20 ml of 0.5% bupivacaine will be injected through the needle.
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Ultrasound Guided Combined Rhomboid Intercostal Sub-serratus Plane Blocks — Ultrasound Guided Combined Rhomboid Intercostal Sub-serratus Plane Blocks
  Arms: Ultrasound guided Rhomboid intercostal block sub-serratus plane block (RISS).
Procedure: Erector Spinae Plane Block — Erector Spinae Plane Block
  Arms: Ultrasound guided Erector spinae plane block (ESPB)

SUMMARY:
Acute post-mastectomy pain can cause adverse impacts on the patients as delayed discharge from post-operative recovery area, impairs pulmonary and immune functions, increases risk of ileus, thromboembolism, myocardial infarction and may lead to increased length of hospital stay. It is also an important factor leading to the development of chronic post mastectomy pain syndrome (PMPS) in almost half of the patients.

Various regional anesthetic techniques have been described for postoperative pain relief after mastectomy, for example, thoracic epidural anesthesia, intercostal nerve block, paravertebral block, serratus anterior plane block, and pectoral nerve I and II blocks. All of them offer satisfactory pain relief after mastectomy.

Erector spinae plane block is a novel para-spinal regional anesthesia technique, , promises to provide effective visceral as well as somatic analgesia after carcinoma of the breast surgeries.

The ultrasound-guided rhomboid intercostal block sub-serratus plane block (RISS) is a novel analgesic technique The RISS block anesthetizes the lateral cutaneous branches of the thoracic intercostal nerves and can be used in multiple clinical settings for chest wall and upper abdominal analgesia

DETAILED DESCRIPTION:
Breast cancer is the most common diagnosed malignancy among females and the 5th cause of cancer-related deaths with an estimated number of 2.3 million new cases and 685,000 deaths worldwide in 2020.

Different modalities are used for management of breast cancer including surgery, radiation therapy (RT), chemotherapy (CT), endocrine (hormone) therapy (ET), and targeted therapy. Modified Radical Mastectomy (MRM) is one of the main modalities of breast cancer treatment. It accounts for 31% of all breast surgeries. It has been reported that 40% of the females complain from moderate-to-severe pain in the immediate post-operative period after breast cancer surgery.

Acute post-mastectomy pain can cause adverse impacts on the patients as delayed discharge from post-operative recovery area, impairs pulmonary and immune functions, increases risk of ileus, thromboembolism, myocardial infarction and may lead to increased length of hospital stay. It is also an important factor leading to the development of chronic post mastectomy pain syndrome (PMPS) in almost half of the patients.

Various regional anesthetic techniques have been described for postoperative pain relief after mastectomy, for example, thoracic epidural anesthesia, intercostal nerve block, paravertebral block, serratus anterior plane block, and pectoral nerve I and II blocks. All of them offer satisfactory pain relief after mastectomy.

Erector spinae plane block is a novel para-spinal regional anesthesia technique, promises to provide effective visceral as well as somatic analgesia after carcinoma of the breast surgeries.

The ultrasound-guided rhomboid intercostal block (RIB) and rhomboid intercostal block sub-serratus plane block (RISS) are two novel analgesic techniques . Additionally, the RISS block anesthetizes the lateral cutaneous branches of the thoracic intercostal nerves and can be used in multiple clinical settings for chest wall and upper abdominal analgesia

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer female patients.
2. ASA class II and III.
3. Age ≥ 18 and ≤ 60 Years.
4. Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.
5. Type of surgery; elective breast cancer surgery (either modified radical mastectomy or conservative breast surgery) combined with axillary dissection.

Exclusion Criteria:

1. Patient refusal.
2. Age <18 years or >65 years.
3. BMI <20 kg/m2 and >35 kg/m2.
4. Major medical conditions.
5. Pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Total post-operative morphine consumption. | 24 hours after the surgery
  The total 24-hour morphine consumption will be recorded for every patient post operative.

SECONDARY OUTCOMES:
Total intra-operative fentanyl consumption | 2-3 hours (Surgery time) surgery
  the rescue analgesia will be administered intra-operative by fentanyl IV and the total fentanyl used will be recorded and compared between the groups
1st time opioids requested post-operative. | 24 hours after the surgery
  In case of postoperative pain recorded, rescue analgesia will be provided as IV morphine (3 mg) then continuous infusion of morphine through Patient Controlled Analgesia ( PCA ) to keep the VAS scores<3. The total 24-hour morphine consumption will be recorded for every patient.
Changes and stability in Mean Arterial Blood Pressure (MAP) | every 15 minutes during the surgery then at 1, 2, 4, 8, 12, 16, 20 and 24 hours postoperatively
  Change in Mean Arterial Blood Pressure (MAP) in mmHg
Changes and stability in Heart Rate (HR) | every 15 minutes during the surgery then at 1, 2, 4, 8, 12, 16, 20 and 24 hours postoperatively
  Change in heart rate (HR) in beat\min

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Sharawy Abdelrahman Aboul Nasr, MD, Principal Investigator — National Cancer Institute Cairo University
Locations (1):
- National Cancer Institute - Cairo University, Cairo, Egypt